CLINICAL TRIAL: NCT00593203
Title: Molecular Neurosurgical Tissue Bank
Brief Title: Brain Tissue Specimen Collection
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Reid Thompson, Director, Vanderbilt University Medical Center
Other Study IDs: 030372
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain Tissue, blood and cerebral spinal fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The Molecular Neurosurgical Tissue Bank will function as a tissue or specimen repository for biopsy specimens from patients (both adult and pediatric) undergoing brain surgery and brain procedures.

DETAILED DESCRIPTION:
The Molecular Neurosurgical Tissue Bank will function as a tissue or specimen repository for biopsy specimens from patients (both adult and pediatric) undergoing brain surgery and brain procedures. Leftover tissue removed during the course of brain surgery will be collected and stored in neurosurgical laboratories for use in medical research that might be currently ongoing or for future research. In addition, blood and cerebral spinal fluid samples will also be collected and stored. Leftover cerebral spinal fluid (CSF) will be collected during standard of care procedures (lumbar punctures or ventricular drains) that take place at time of diagnosis, completion of therapy and relapse of disease or during neurosurgery. Blood will be drawn at time of routine lab draws required during the surgery or procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having any type of brain surgery, where a specimen will be collected.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: infant through Adults
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2003-05; Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Reid C. Thompson, M.D., Principal Investigator — Vanderbilt University Medical Center, Department of Neurological Surgery
Locations (1):
- Vanderbilt University Medical Center, Deptartment of Neurological Surgery, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No